CLINICAL TRIAL: NCT04197258
Title: Evaluation of the Impact of an Individual Peer Support Intervention for Stroke Patients When Returning Home: a Mixed Methods Pilot Study
Acronym: PARADE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 69HCL19_0233
Record Dates: First submitted 2019-12-05; First posted 2019-12-13 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Stroke
Keywords: Stroke; Peer support
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention group (Experimental): For 6 months after discharge, patients in the intervention group will benefit from peer support by a trained patient (number and frequency of contacts defined according to the patient's needs).
  The intervention aims to improve the patient's ability to manage his or her situation and meet his or her needs upon discharge at home, including identifying and seeking for the necessary health or social resources
  Interventions: Other: Peer support
- control group (No Intervention): Patients included in the control group before intervention will receive the usual practices. As part of the study, they will be contacted for data collection 6 months after the transition to home by a clinical research associate.

INTERVENTIONS:
Other: Peer support — The intervention studied is the psycho-social support by a peer-helper to the patients and their main informal caregiver during the return home following a stay in rehabilitation center for a stroke.
  Peer support intervention will be based on evidence, Bandura's social learning and social support theory, and the results of our ongoing study of the needs of patients and their caregivers as a result of returning home (Stroke69). It will include a meeting before the discharge and a regular follow-up for 6 months (face-to-face meetings, virtual or by phone), adapted to the needs of the patient and his caregiver, taking into account the social environment and in connection with the devices existing sanitary and social.
  Arms: intervention group

SUMMARY:
Going back home following a stroke is a key step for the patient and his or her relatives. Due to the brutality of stroke and increasingly shorter in-hospital lengths of stay, patients and their families must adapt quickly to the patient's new health functioning and the new caregiving and support role for family members.

Peer support could be an innovative and inexpensive approach to addressing these issues. Peer-helpers are patient-partners who put their experiential knowledge from life with the disease at the disposal of other patients to offer them social and emotional support in the management of the disease in connection with care, social and community structures. Group peer support programs face organizational challenges and fail to address the full range of patient needs for stroke home visits. Individualized and more flexible support could better meet the needs of patients. Our hypothesis is that individual peer support improves quality of life and patient empowerment during the discharge period compared to usual practice.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient,
* Having had a first confirmed, ischemic or hemorrhagic stroke
* Managed in the participating rehabilitation center
* Whose discharge to home directly from the rehabilitation center is planned
* Presenting a modified Rankin score of 1 to 3 when deciding to leave the stroke center
* Having given its written consent
* Whose main residence is located in the Rhône department
* Aphasic patients may be included if a caregiver can follow up with the case manager

Exclusion Criteria:

* Patient living in an institution prior to stroke
* included in a gerontological network before stroke
* Patient unable to understand quality of life questionnaires
* Patient with unstable medical or psychological conditions who, in the opinion of the investigator, could lead the subject to be non-compliant or uncooperative during the study or could compromise patient safety or participation in the study
* Patient under guardianship or curatorship
* Patient not affiliated to a social health insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-10-09 (Actual); Primary Completion 2026-12-05 (Estimated); Study Completion 2026-12-05 (Estimated)

PRIMARY OUTCOMES:
Feasibility measure | 6 months
  The feasibility of the intervention will be evaluated as success with a combined criteria including:
  * Recruitment and training of 2 peer helpers,
  * Support offered to 20 patients by the peer helpers during the intervention period defined by at least one meeting before and one contact after discharge per patient included in period after,
  * Good acceptability by patients, carers and peer helpers. These data will be collected by a qualitative approach associating semi-directive interviews, focus groups and participant observation.

SECONDARY OUTCOMES:
Quality of life between the discharge from hospital and 6 months | 6 months
  Evolution of the dimensions of the SIS at hospital discharge and 6 months: force dimension
Quality of life between the discharge from hospital and 6 months | 6 months
  Evolution of the dimensions of the SIS at hospital discharge and 6 months: manual function
Quality of life between the discharge from hospital and 6 months | 6 months
  Evolution of the dimensions of the SIS at hospital discharge and 6 months: AVQ/AVD
Quality of life between the discharge from hospital and 6 months | 6 months
  Evolution of the dimensions of the SIS at hospital discharge and 6 months: Mobility
Quality of life between the discharge from hospital and 6 months | 6 months
  Evolution of the dimensions of the SIS at hospital discharge and 6 months: Communication and Emotions
Quality of life between the discharge from hospital and 6 months | 6 months
  Evolution of the dimensions of the SIS at hospital discharge and 6 months: Memory and thinking
Quality of life between the discharge from hospital and 6 months | 6 months
  Evolution of the dimensions of the SIS at hospital discharge and 6 months: global recovery
Anxiety and depression scores between discharge and 6 months | 6 months
  Evolution of anxiety and depression scores between discharge and 6 months after discharge, measured by the Hospital Anxiety and Depression scale (HADS) score
Patient activation Measure | 6 months
  Evolution of patient activation between discharge and 6 months after discharge, measured by the Patient activation Measure (PAM) score
Disability | 6 months
  proportion of patients with disabilities at 6 months evaluated by the Modified Rankin Scale (no disability corresponding to mRs<3)
Adherence | 6 months
  proportion of adherent patients at 6 months evaluated by the Medication Adherence Rating Scale (MARS)
Human, material and financial assistance provided at home | 6 months
  Human, material and financial assistance provided at home collected by interviewing the patient
Satisfaction measure | 6 months
  Perceived satisfaction of the support received on during the discharge period will be collected by interviewing the patient
Caregiver burden | 6 months
  Evolution of caregiver burden between discharge and 6 months after discharge, measured by the Zarit burden scale
Caregiver satisfaction | 6 months
  Perceived caregiver satisfaction of the support during the patient's discharge period will be collected by interviewing caregiver

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Henry Gabrielle, Saint-Genis-Laval, France